CLINICAL TRIAL: NCT02601859
Title: Evaluation of Lithium as a Glycogen-Synthase-Kinase-3 (GSK-3) Inhibitor in Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2014MH08
Record Dates: First submitted 2015-11-02; First posted 2015-11-10 (Estimated); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Lithium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phase 3 (Experimental): Administration of Lithium to 11 individuals with MCI (non-randomised) for 9 weeks. Lithium dose escalates from 100mg to 200mg to 400mg, then a 3 week wash out period, total study duration 12 weeks. Blood samples taken at regular intervals throughout trial and analysed for GSK-3 enzyme activity in blood.
  Interventions: Drug: Lithium Carbonate

INTERVENTIONS:
Drug: Lithium Carbonate

SUMMARY:
The project is designed to generate critical information to design and justify a robust trial on lithium prevention of the onset of Alzheimer's disease (AD). Lithium exerts and inhibitory effect on Glycogen synthase kinase 3 (GSK-3) a brain biomarker of neuroprotection. The study consists of 3 phases:

1. Phase 1 investigates rats to establish a reliable method to measure brain biomarker activity levels from blood biomarker activity.
2. Phase 2 will determine whether the GSK3 enzyme activity is significantly different in subjects with MCI compared to normal individuals.
3. Phase 3 investigates patients with MCI taking lithium to establish the minimum lithium dose required to inhibit the activity of GSK-3.

DETAILED DESCRIPTION:
Lithium has been used for decades to treat Bipolar Affective Disorder. Some of its therapeutic benefits are through the inhibition of the enzyme Glycogen Synthase Kinase-3 (GSK-3). GSK3 activity is associated with the development of several aspects of AD and thus lithium can regulate an enzyme linked to AD development. As an important step towards designing a clinical trial to investigate the potential of lithium for AD prevention the investigators propose to establish the minimum dose of lithium needed to block GSK3 in people with Mild Cognitive Impairment (MCI), a high-risk condition for progression to AD. The study will establish whether GSK3 activity is altered in MCI and monitor lithium regulation of GSK3 biomarkers in this population. At the same time the study will investigate how GSK3 measured in blood relates to GSK3 activity in the brain in a small animal study. In further preparation for a future large scale trial, this pilot study will generate technical data to develop the technique of using Magnetic Resonance Spectroscopy (MRS) as a biomarker to detect the earliest brain changes of AD.

Recruitment will be shared between the two sites for this study, Dundee and Oxford. The study will involve 12 patients with MCI and 12 controls, who will be asked for two sets of blood tests, and 20 patients with MCI who consent to take Lithium who will be asked for blood tests at regular intervals. For all participants the study period is 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Mild Cognitive Impairment (MCI).

Exclusion Criteria:

* Previous hypersensitivity to Lithium or other contraindication to Lithium carbonate Priadel (see most recent SmPC), Dementia Diabetes BMI <18 or >30 Rheumatoid Arthritis and Autoimmune Inflammatory disorders Currently taking NSAIDS Moderate renal failure (defined in BNF by gGFR <60 mL/minute/1.73m2) or severe Renal failure (defined in BNF by eGFR <29 mL/minute/1.73m2 Addison's disease, Brugada syndrome (or family history of Brugada syndrome), cardiac insufficiency, congestive cardiac failure, epilepsy, suicidality incapacity to consent currently prescribed lithium participation in another clinical trial of an Investigational Medicinal Product (IMP) in the last 28 days.

Uncontrolled serious concomitant physical illness

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-08; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
GSK-3 activity in PBMC isolates | 12 weeks
  Measures are six robust measures are of upstream/downstream signalling and GSK3 function and will be validated by other work by the investigators. GSK-3 function will be described according to plasma Lithium concentration.

REFERENCES:
- [Result] Duthie A, van Aalten L, MacDonald C, McNeilly A, Gallagher J, Geddes J, Lovestone S, Sutherland C. Recruitment, Retainment, and Biomarkers of Response; A Pilot Trial of Lithium in Humans With Mild Cognitive Impairment. Front Mol Neurosci. 2019 Jun 28;12:163. doi: 10.3389/fnmol.2019.00163. eCollection 2019. PMID 31316348